CLINICAL TRIAL: NCT00986232
Title: A Dose Selection Study in Healthy Children Comparing Measles Mumps, Rubella, and Varicella (ProQuad) Vaccine to M-M-R II Given Concomitantly With Process Upgrade Varicella Vaccine (PUVV) in Separate Injections
Brief Title: ProQuad Dose Selection Study (V221-011)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V221-011; 2009_667
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Results first posted 2010-02-15 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): ProQuad (low dose)
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live
- 2 (Experimental): ProQuad (middle dose)
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live
- 3 (Experimental): ProQuad (high dose)
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live
- 4 (Active Comparator): M-M-R II + PUVV
  Interventions: Biological: Comparator: M-M-R II; Biological: Comparator: PUVV

INTERVENTIONS:
Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live — a single 0.5 mL subcutaneous injection of ProQuad (low, middle, or high dose) at Day 0 and Day 90
  Other Names: ProQuad
  Arms: 1; 2; 3
Biological: Comparator: M-M-R II — A single 0.5 mL subcutaneous injection at Day 0
  Arms: 4
Biological: Comparator: PUVV — A single 0.5 mL subcutaneous injection at Day 0
  Arms: 4

SUMMARY:
A Study comparing three different doses of ProQuad to concomitant administration of M-M-R II and PUVV (Process Upgrade Varicella Vaccine) vaccines.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Negative clinical history of measles, mumps, rubella, varicella, and zoster

Exclusion Criteria:

* Previous receipt of measles, mumps, rubella and/or varicella vaccine either alone or in combination
* Any immune impairment or deficiency
* Exposure to measles, mumps, rubella, varicella, or zoster in the 4 weeks prior to vaccination
* Vaccination with an inactive vaccine with in the past 14 days
* Vaccination with a live vaccine within the past 30 days
* Immune globulin or any blood product administered in the past 3 months

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1551 (Actual)
Dates: Start 1999-04; Primary Completion 2000-04 (Actual); Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Shinefield H, Black S, Williams WR, Marchant C, Reisinger K, Stewart T, Meissner HC, Guerrero J, Klopfer SO, Xu J, Schodel F, Kuter BJ; Dose Selection Study Group for Proquad. Dose-response study of a quadrivalent measles, mumps, rubella and varicella vaccine in healthy children. Pediatr Infect Dis J. 2005 Aug;24(8):670-5. doi: 10.1097/01.inf.0000172901.29621.e9. PMID 16094218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 clinical sites in the United States
  Date first participant visit: 08-Apr-1999
  Date last participant visit: 03-Apr-2000
Groups:
- ProQuad™ (Low Dose): One ProQuad™ (3.48 log10 plaque-forming units [PFU]/0.5-mL dose) subcutaneous (SQ) injection administered on Day 0, followed by a second injection of the same material approximately 90 days later.
- ProQuad™ (Middle Dose): One ProQuad™ (3.97 log10 PFU/0.5-mL dose) SQ injection administered on Day 0, followed by a second injection of the same material approximately 90 days later.
- ProQuad™ (High Dose): One ProQuad™ (4.25 log10 PFU/0.5-mL dose) SQ injection administered on Day 0, followed by a second injection of the same material approximately 90 days later.
- M-M-R™ II + PUVV (Process Upgrade Varicella Vaccine): One M-M-R™ II (0.5-mL) SQ injection administered concomitantly with one PUVV (0.5-mL) SQ injection, at separate injection sites, on Day 0.
Period: Overall Study
Arm/Group | ProQuad™ (Low Dose) | ProQuad™ (Middle Dose) | ProQuad™ (High Dose) | M-M-R™ II + PUVV (Process Upgrade Varicella Vaccine)
Started | 387 | 393 (Excludes 1 patient who was randomized to receive ProQuad (Middle Dose), but was not vaccinated.) | 381 | 390 (Excludes 1 patient who was randomized to receive M-M-R™ II + PUVV, but was not vaccinated.)
Vaccination Visit 1 | 387 | 393 | 381 | 390
Vaccination Visit 2 | 360 | 365 | 360 | 0
Completed | 336 | 343 | 346 | 370
Not Completed | 51 | 50 | 35 | 20
Not completed — Adverse Event | 1 | 2 | 3 | 0
Not completed — Lost to Follow-up | 19 | 12 | 12 | 7
Not completed — Protocol Violation | 2 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 13 | 16 | 12 | 3
Not completed — Missed one or more bleeds | 13 | 10 | 6 | 7
Not completed — Incomplete safety follow-up | 3 | 7 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ProQuad™ (Low Dose) | ProQuad™ (Middle Dose) | ProQuad™ (High Dose) | M-M-R™ II + PUVV (Process Upgrade Varicella Vaccine) | Total
Number analyzed (Participants) | 387 | 393 | 381 | 390 | 1551
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.9 (1.5) | 12.9 (1.5) | 12.9 (1.5) | 13.0 (1.7) | 12.9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 181 | 192 | 161 | 720
  Male | 201 | 212 | 189 | 229 | 831
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 65 | 55 | 64 | 54 | 238
  Asian/Pacific | 19 | 11 | 19 | 13 | 62
  Caucasian | 241 | 267 | 251 | 262 | 1021
  Hispanic | 34 | 44 | 22 | 25 | 125
  Native American | 1 | 1 | 1 | 0 | 3
  Other | 27 | 15 | 24 | 36 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Varicella Glycoprotein Enzyme-Linked Immunosorbent Assay (gpELISA) Antibody Titer ≥ 5 gpELISA Units
Description: Antibody response to Varicella at 6 weeks postvaccination in participants with baseline titer <1.25 gpELISA units
Time Frame: 6 weeks postvaccination
Population: The per-protocol analysis set included participants who had pre- and post-randomization blood samples within predefined day ranges, were seronegative to varicella at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Groups:
- ProQuad™ (Low Dose) After 1 Injection; ProQuad™ (Low Dose) After 2 Injections: One ProQuad™ (3.48 log10 plaque-forming units [PFU]/0.5-mL dose) subcutaneous (SQ) injection administered on Day 0, followed by a second injection of the same material approximately 90 days later.
- ProQuad™ (Middle Dose) After 1 Injection; ProQuad™ (Middle Dose) After 2 Injections: One ProQuad™ (3.97 log10 PFU/0.5-mL dose) SQ injection administered on Day 0, followed by a second injection of the same material approximately 90 days later.
- ProQuad™ (High Dose) After 1 Injection; ProQuad™ (High Dose) After 2 Injections: One ProQuad™ (4.25 log10 PFU/0.5-mL dose) SQ injection administered on Day 0, followed by a second injection of the same material approximately 90 days later.
- M-M-R™ II + PUVV After 1 Injection: One M-M-R™ II (0.5-mL) SQ injection administered concomitantly with one PUVV (0.5-mL) SQ injection, at separate injection sites, on Day 0.
Arm/Group | ProQuad™ (Low Dose) After 1 Injection | ProQuad™ (Low Dose) After 2 Injections | ProQuad™ (Middle Dose) After 1 Injection | ProQuad™ (Middle Dose) After 2 Injections | ProQuad™ (High Dose) After 1 Injection | ProQuad™ (High Dose) After 2 Injections | M-M-R™ II + PUVV After 1 Injection
Number analyzed (Participants) | 310 | 300 | 313 | 303 | 307 | 309 | 320
Participants | 198 | 299 | 253 | 303 | 272 | 306 | 298

2. Secondary Outcome: Number of Participants With Postvaccination Measles Enzyme-Linked Immunosorbent Assay (ELISA) Antibody Titer ≥ 207.5 mIU/mL
Description: Antibody response to measles at 6 weeks postvaccination in participants initially seronegative (a titer <207.5 mIU/mL) to measles at baseline
Time Frame: 6 weeks postvaccination
Population: The per-protocol analysis set included participants who had pre- and post-randomization blood samples within predefined day ranges, were seronegative to measles at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™ (Low Dose) After 1 Injection | ProQuad™ (Low Dose) After 2 Injections | ProQuad™ (Middle Dose) After 1 Injection | ProQuad™ (Middle Dose) After 2 Injections | ProQuad™ (High Dose) After 1 Injection | ProQuad™ (High Dose) After 2 Injections | M-M-R™ II + PUVV After 1 Injection
Number analyzed (Participants) | 324 | 313 | 342 | 328 | 323 | 326 | 350
Participants | 321 | 311 | 338 | 327 | 321 | 326 | 349

3. Secondary Outcome: Number of Participants With Postvaccination Mumps ELISA Antibody Titer ≥ 2.0 Ab Units/mL
Description: Antibody response to Mumps at 6 weeks postvaccination in participants initially seronegative (a titer < 2.0 Ab units/mL) to Mumps at baseline
Time Frame: 6 weeks Postvaccination
Population: The per-protocol analysis set included participants who had pre- and post-randomization blood samples within predefined day ranges, were seronegative to mumps at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™ (Low Dose) After 1 Injection | ProQuad™ (Low Dose) After 2 Injections | ProQuad™ (Middle Dose) After 1 Injection | ProQuad™ (Middle Dose) After 2 Injections | ProQuad™ (High Dose) After 1 Injection | ProQuad™ (High Dose) After 2 Injections | M-M-R™ II + PUVV After 1 Injection
Number analyzed (Participants) | 334 | 322 | 347 | 331 | 331 | 335 | 351
Participants | 333 | 322 | 344 | 330 | 325 | 335 | 350

4. Secondary Outcome: Number of Participants With Postvaccination Rubella ELISA Antibody Titer ≥ 10 IU/mL
Description: Antibody response to Rubella at 6 weeks postvaccination in participants initially seronegative (a titer <10 IU/mL) to Rubella at baseline
Time Frame: 6 weeks Postvaccination
Population: The per-protocol analysis set included participants who had pre- and post-randomization blood samples within predefined day ranges, were seronegative to rubella at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™ (Low Dose) After 1 Injection | ProQuad™ (Low Dose) After 2 Injections | ProQuad™ (Middle Dose) After 1 Injection | ProQuad™ (Middle Dose) After 2 Injections | ProQuad™ (High Dose) After 1 Injection | ProQuad™ (High Dose) After 2 Injections | M-M-R™ II + PUVV After 1 Injection
Number analyzed (Participants) | 335 | 319 | 347 | 333 | 333 | 335 | 357
Participants | 335 | 319 | 343 | 332 | 326 | 335 | 352

5. Secondary Outcome: Number of Participants With Serious Vaccine-Related Clinical Adverse Experiences (CAEs)
Description: Participants with a serious vaccine-related CAE (an AE which is assessed by an investigator/qualified physician as being related to study vaccine and results in death, persistent or significant disability/incapacity, prolongs an existing inpatient hospitalization, is life-threatening, a congenital anomaly/birth defect, a cancer, or an overdose).
Time Frame: 6 weeks Postvaccination Visit 1 or Visit 2
Population: All participants with follow-up for safety were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | ProQuad™ (Low Dose) After 1 Injection | ProQuad™ (Low Dose) After 2 Injections | ProQuad™ (Middle Dose) After 1 Injection | ProQuad™ (Middle Dose) After 2 Injections | ProQuad™ (High Dose) After 1 Injection | ProQuad™ (High Dose) After 2 Injections | M-M-R™ II + PUVV After 1 Injection
Number analyzed (Participants) | 378 | 353 | 387 | 361 | 377 | 358 | 381
Participants
  With Serious Vaccine-Related CAEs | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Without Serious Vaccine-Related CAEs | 378 | 353 | 386 | 361 | 377 | 358 | 381

6. Secondary Outcome: Antibody Response to Varicella at 6 Weeks Postvaccination in Participants With Baseline Titer < 1.25 gpELISA Units - Geometric Mean Titer (GMT)
Description: Postvaccination observed Geometric Mean Titer (GMT) of Varicella antibody. (Titers measured using Varicella zoster virus (VZV) gpELISA.)
Time Frame: 6 weeks Postvaccination
Population: The per-protocol analysis set included participants who had pre- and post-randomization blood samples within predefined day ranges and followed protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | ProQuad™ (Low Dose) After 1 Injection | ProQuad™ (Low Dose) After 2 Injections | ProQuad™ (Middle Dose) After 1 Injection | ProQuad™ (Middle Dose) After 2 Injections | ProQuad™ (High Dose) After 1 Injection | ProQuad™ (High Dose) After 2 Injections | M-M-R™ II + PUVV After 1 Injection
Number analyzed (Participants) | 310 | 300 | 313 | 303 | 307 | 309 | 320
mcg/mL | 5.7 [5.0 to 6.5] | 167.7 [145.6 to 193.2] | 10.5 [9.4 to 11.7] | 381.0 [335.8 to 432.4] | 11.9 [10.8 to 13.1] | 469.4 [405.5 to 543.4] | 16.5 [15.1 to 18.1]

7. Secondary Outcome: Antibody Response to Measles at 6 Weeks Postvaccination in Participants Initially Seronegative to Measles at Baseline - Geometric Mean Titer (GMT)
Description: Postvaccination observed Geometric Mean Titer (GMT) of Measles antibody. (Titers measured using Measles ELISA.)
Time Frame: 6 weeks Postvaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | ProQuad™ (Low Dose) After 1 Injection | ProQuad™ (Low Dose) After 2 Injections | ProQuad™ (Middle Dose) After 1 Injection | ProQuad™ (Middle Dose) After 2 Injections | ProQuad™ (High Dose) After 1 Injection | ProQuad™ (High Dose) After 2 Injections | M-M-R™ II + PUVV After 1 Injection
Number analyzed (Participants) | 324 | 313 | 342 | 328 | 323 | 326 | 350
mcg/mL | 251.8 [229.9 to 275.8] | 549.7 [484.8 to 623.4] | 309.5 [280.8 to 341.3] | 783.0 [681.8 to 899.1] | 315.4 [286.4 to 347.3] | 747.9 [656.9 to 851.7] | 253.5 [230.5 to 278.8]

8. Secondary Outcome: Antibody Response to Mumps at 6 Weeks Postvaccination in Participants Initially Seronegative to Mumps at Baseline - Geometric Mean Titer (GMT)
Description: Postvaccination observed Geometric Mean Titer (GMT) of Mumps antibody. (Titer measured using Mumps ELISA.)
Time Frame: 6 weeks Postvaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | ProQuad™ (Low Dose) After 1 Injection | ProQuad™ (Low Dose) After 2 Injections | ProQuad™ (Middle Dose) After 1 Injection | ProQuad™ (Middle Dose) After 2 Injections | ProQuad™ (High Dose) After 1 Injection | ProQuad™ (High Dose) After 2 Injections | M-M-R™ II + PUVV After 1 Injection
Number analyzed (Participants) | 334 | 322 | 347 | 331 | 331 | 335 | 351
mcg/mL | 102.0 [90.0 to 115.7] | 277.7 [252.0 to 305.9] | 106.3 [94.4 to 119.8] | 244.1 [220.3 to 270.3] | 114.7 [101.3 to 130.0] | 286.0 [259.2 to 315.7] | 97.4 [87.5 to 108.5]

9. Secondary Outcome: Antibody Response to Rubella at 6 Weeks Postvaccination in Participants Initially Seronegative to Rubella at Baseline - Geometric Mean Titer (GMT)
Description: Postvaccination observed Geometric Mean Titer (GMT) of Rubella antibody. (Titers measured using Rubella ELISA.)
Time Frame: 6 weeks postvaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | ProQuad™ (Low Dose) After 1 Injection | ProQuad™ (Low Dose) After 2 Injections | ProQuad™ (Middle Dose) After 1 Injection | ProQuad™ (Middle Dose) After 2 Injections | ProQuad™ (High Dose) After 1 Injection | ProQuad™ (High Dose) After 2 Injections | M-M-R™ II + PUVV After 1 Injection
Number analyzed (Participants) | 335 | 319 | 347 | 333 | 333 | 335 | 357
mcg/mL | 131.4 [119.6 to 144.5] | 263.7 [239.0 to 291.0] | 122.5 [110.7 to 135.5] | 230.7 [207.8 to 256.0] | 115.5 [104.9 to 127.2] | 254.2 [230.5 to 280.3] | 128.5 [116.5 to 141.7]

ADVERSE EVENTS:
Time Frame: Participants were followed for safety for 42 days after each scheduled vaccination.
Description: Number of participants reported as "At Risk" is the number of participants with follow-up.
Groups:
- ProQuad (Low Dose) After Injection 1; ProQuad (Low Dose) After Injection 2: One ProQuad™ (3.48 log10 plaque-forming units [PFU]/0.5-mL dose) subcutaneous (SQ) injection administered on Day 0, followed by a second injection of the same material approximately 90 days later.
- ProQuad (Middle Dose) After Injection 1; ProQuad (Middle Dose) After Injection 2: One ProQuad™ (3.97 log10 PFU/0.5-mL dose) SQ injection administered on Day 0, followed by a second injection of the same material approximately 90 days later.
- ProQuad (High Dose) After Injection 1; ProQuad (High Dose) After Injection 2: One ProQuad™ (4.25 log10 PFU/0.5-mL dose) SQ injection administered on Day 0, followed by a second injection of the same material approximately 90 days later.
Arm/Group | ProQuad (Low Dose) After Injection 1 | ProQuad (Middle Dose) After Injection 1 | ProQuad (High Dose) After Injection 1 | M-M-R™ II + PUVV (Process Upgrade Varicella Vaccine) | ProQuad (Low Dose) After Injection 2 | ProQuad (Middle Dose) After Injection 2 | ProQuad (High Dose) After Injection 2
Serious Adverse Events (participants affected / at risk) | 2/378 | 3/387 | 1/377 | 1/381 | 1/353 | 0/361 | 2/358
Other Adverse Events (participants affected / at risk) | 286/378 | 286/387 | 289/377 | 297/381 | 253/353 | 258/361 | 254/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ProQuad (Low Dose) After Injection 1 (N=378) | ProQuad (Middle Dose) After Injection 1 (N=387) | ProQuad (High Dose) After Injection 1 (N=377) | M-M-R™ II + PUVV (Process Upgrade Varicella Vaccine) (N=381) | ProQuad (Low Dose) After Injection 2 (N=353) | ProQuad (Middle Dose) After Injection 2 (N=361) | ProQuad (High Dose) After Injection 2 (N=358)
Bacteremia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Seizure, febrile (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Laryngotracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory distress, newborn (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Otitis media (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ProQuad (Low Dose) After Injection 1 (N=378) | ProQuad (Middle Dose) After Injection 1 (N=387) | ProQuad (High Dose) After Injection 1 (N=377) | M-M-R™ II + PUVV (Process Upgrade Varicella Vaccine) (N=381) | ProQuad (Low Dose) After Injection 2 (N=353) | ProQuad (Middle Dose) After Injection 2 (N=361) | ProQuad (High Dose) After Injection 2 (N=358)
Asthenia/Fatigue (General disorders) | 2 | 1 | 4 | 2 | 1 | 1 | 0
Candidiasis (General disorders) | 1 | 1 | 4 | 2 | 4 | 1 | 2
Fever (General disorders) | 116 | 128 | 145 | 136 | 81 | 98 | 99
Infection, Viral (Infections and infestations) | 12 | 16 | 16 | 14 | 10 | 11 | 14
Malaise (General disorders) | 4 | 2 | 4 | 1 | 2 | 0 | 2
Trauma (Injury, poisoning and procedural complications) | 4 | 8 | 1 | 4 | 2 | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 8 | 10 | 6 | 6 | 3 | 6 | 1
Candidiasis, Oral (Gastrointestinal disorders) | 4 | 1 | 1 | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 6 | 2 | 2 | 2 | 3 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 34 | 23 | 31 | 31 | 19 | 26 | 16
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 0 | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 3 | 4 | 5 | 5 | 4 | 5
Gastroenteritis, Infectious (Gastrointestinal disorders) | 8 | 4 | 5 | 2 | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 12 | 16 | 21 | 23 | 19 | 17 | 23
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 4 | 0 | 0 | 0 | 0
Allergy (Immune system disorders) | 4 | 4 | 3 | 3 | 1 | 4 | 2
Crying (Nervous system disorders) | 4 | 4 | 1 | 3 | 2 | 0 | 3
Irritability (Psychiatric disorders) | 52 | 49 | 51 | 42 | 29 | 28 | 29
Somnolence (Psychiatric disorders) | 4 | 1 | 1 | 1 | 0 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 3 | 4 | 6 | 6 | 13
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1 | 1 | 1 | 2 | 4
Congestion, Nasal (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 9 | 5 | 6 | 3 | 6
Congestion, Respiratory (Respiratory, thoracic and mediastinal disorders) | 6 | 14 | 7 | 8 | 13 | 20 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 20 | 20 | 25 | 26 | 33 | 32
Infection, Respiratory, Upper (Infections and infestations) | 60 | 58 | 67 | 64 | 82 | 110 | 93
Influenza (Infections and infestations) | 0 | 0 | 3 | 1 | 5 | 2 | 5
Laryngotracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 8 | 4 | 8 | 6 | 7
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 10 | 13 | 7 | 6 | 11
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 3 | 0 | 3 | 4
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2 | 1 | 2 | 3 | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 28 | 34 | 38 | 41 | 28 | 29 | 27
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3 | 5 | 8 | 7 | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 0 | 5 | 4 | 4 | 4
Bite/Sting, Non-Venomous (Injury, poisoning and procedural complications) | 4 | 9 | 4 | 4 | 1 | 1 | 3
Burn (Injury, poisoning and procedural complications) | 0 | 2 | 4 | 0 | 3 | 0 | 0
Dermatitis, Contact (Skin and subcutaneous tissue disorders) | 6 | 3 | 7 | 4 | 2 | 4 | 1
Eczema (Skin and subcutaneous tissue disorders) | 7 | 6 | 4 | 4 | 4 | 4 | 2
Miliaria Rubra (Skin and subcutaneous tissue disorders) | 10 | 9 | 11 | 7 | 3 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 15 | 11 | 19 | 7 | 13 | 12
Rash, Diaper (Skin and subcutaneous tissue disorders) | 16 | 8 | 8 | 14 | 6 | 7 | 7
Rash, Measles/Rubella-Like (Skin and subcutaneous tissue disorders) | 13 | 18 | 18 | 14 | 1 | 2 | 1
Rash, Varicella-Like (Skin and subcutaneous tissue disorders) | 8 | 12 | 11 | 8 | 1 | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 0 | 1 | 0 | 4
Viral Exanthema (Infections and infestations) | 14 | 16 | 15 | 18 | 6 | 9 | 6
Conjunctivitis (Eye disorders) | 6 | 10 | 10 | 10 | 5 | 5 | 6
Otitis (Ear and labyrinth disorders) | 10 | 7 | 6 | 5 | 10 | 3 | 7
Otitis Media (Ear and labyrinth disorders) | 34 | 37 | 34 | 42 | 53 | 48 | 59
Otitis Media, Serous (Ear and labyrinth disorders) | 4 | 2 | 1 | 3 | 6 | 0 | 1
Pain, Ear (Ear and labyrinth disorders) | 4 | 2 | 2 | 3 | 3 | 3 | 4
Ecchymosis (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 4 | 8 | 4 | 0/0 | 4 | 4 | 2
Erythema (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 48 | 43 | 32 | 0/0 | 36 | 46 | 38
Pain/Tenderness/Soreness (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 84 | 70 | 78 | 0/0 | 57 | 52 | 51
Rash (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 7 | 5 | 7 | 0/0 | 2 | 1 | 2
Swelling (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 29 | 23 | 30 | 0/0 | 31 | 22 | 21
Ecchymosis (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 5 | 0/0 | 0/0 | 0/0
Erythema (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 56 | 0/0 | 0/0 | 0/0
Pain/Tenderness/Soreness (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 90 | 0/0 | 0/0 | 0/0
Swelling (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 36 | 0/0 | 0/0 | 0/0
Ecchymosis (PUVV Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 8 | 0/0 | 0/0 | 0/0
Erythema (PUVV Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 48 | 0/0 | 0/0 | 0/0
Pain/Tenderness/Soreness (PUVV Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 85 | 0/0 | 0/0 | 0/0
Rash (PUVV Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 7 | 0/0 | 0/0 | 0/0
Swelling (PUVV Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 32 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Seven (7) participants received unknown clinical material and 1 participant received diluent only; they were considered to be protocol violators and weren't included in the efficacy/safety analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.